CLINICAL TRIAL: NCT05837494
Title: Comparative Study Between Intra Articular Injection of Ozone With Corticosteroids Versus Plasma Rich in Growth Factors in Limitation of Pain in Knee Osteoarthritis
Brief Title: Intra Articular Injection of Ozone With Corticosteroids vs PRGF in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Hamdy Saied Ayad, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine Faculty Of Medicine Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35293/2/22
Record Dates: First submitted 2023-03-10; First posted 2023-05-01 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Intra Articular Injection; Corticosteroids; Plasma Rich in Growth Factors; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ozone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ozone (Active Comparator)
  Interventions: Drug: Intra-articular Ozone and corticosteroids
- Group PRGF(plasma rich in growth factors) (Active Comparator)
  Interventions: Drug: intra-articular PRGF Method

INTERVENTIONS:
Drug: Intra-articular Ozone and corticosteroids — patients will undergo one session a week for a total of four sessions of intra-articular knee injection with combination of 5ml (25 μg/ml) ozone injection + 2 ml lignocaine 2% + 2 ml Betamethasone sodium phosphate 4 mg.
  Under aseptic precautions. A22-gauge needle was positioned inferior-laterally into the infera-patellar pouch, injection of 2 ml of 4 mg Betamethasone sodium phosphate, and 2 ml injection lignocaine 2% was injected slowly (over 1-2 minutes). The needle was left in space for the 5 ml (25 μg/ml) ozone injection. Patients were advised to avoid strenuous activity for 2-3 days following the intra-articular injection.
  Arms: Group ozone
Drug: intra-articular PRGF Method — Patients will undergoes two doses with 2 weeks interval by injection of already synthetic plasma rich in growth factors [PRGF] vial intra-articularly.
  This vial is formed of lyophilized cake of platelet growth factors in a tightly sealed container stored at 2-8◦C which synthesized under complete aseptic technique by activation of platelets to release its growth factors and cytokines which help in knee cartilage regeneration and act as potent anti-inflammatory to reduce the pain.
  Prior to usage, reconstitution of the product was done using 1 ml saline and 1 ml lignocaine 2% followed by gentle vial rubbing for 3 min then, the mixture was kept at ambient temperature for 5 min to ensure complete protein re-hydration.
  Arms: Group PRGF(plasma rich in growth factors)

SUMMARY:
The aim of this study is to compare the effectiveness of intra-articular injection of ozone with corticosteroids versus plasma rich in growth factors (PRGF) in improvement of pain in knee osteoarthritis patients.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a prevalent degenerative condition in which functional impairment is caused by mechanical and chemical stress against the joint, resulting in pain and decreased range of motion (ROM) .

A multiplicity of treatments has been suggested for this disease : some of which include patient education, medication, exercise prescription, conventional and physical agent modalities such as pulsed radio-frequency, and surgical management , The current therapeutic options available for knee osteoarthritis are not effective and satisfactory for patients, and pain has been complained of by at least 40% of those cases who underwent surgical arthroplasty , Also old age prevalence of knee osteoarthritismake treatment with analgesics has several side effects over stomach, liver and kidney and also surgical one has high morbidities and mortalities for old ages. Therefore, in the last two decades, a large body of work has been performed to develop non-operative or minimally invasive interventions to decrease Knee osteoarthritis symptoms or slow down its progression.

Among These modalities of intra-articular injections the autologous PRP has gained more attention in the treatment of patients with knee osteoarthritis in recent years. Several studies is supporting the use of PRP injection as an effective method for Knee osteoarthritis, as latelet-rich plasma (PRP) could serve as anti-nociceptive and induce cell proliferation. also intra-articular injection of latelet-rich plasma modulates joint environment, promote chondrogenesis and inhibits the destruction of knee joint probably by reducing the production of pro-inflammatory mediators by the supra-physiologic concentrations of biological molecules and growth factors exist in in the granules of the platelets which could potentially reverse the catabolic environment in osteoarthritis, balancing the homeostasis of the joint, and subsequently stimulate the repair of damaged cartilage.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21-65 years
* both genders
* who will be diagnosed with stage 2-3 knee osteoarthritis according to the Kellgren-Lawrence Classification System (K-L) [10], with WOMAC Score > 2 for pain stiffness and physical disabilities
* having symptoms of Knee OA at least 3 months after getting usual conservative treatment like oral analgesics and Therapeutic Exercises.

Exclusion Criteria:

* Patient refusal.
* Patients who will be diagnosed with Stage 1or 4 OA according to K-L Classification
* History of knee trauma within the past month
* History of malignancies
* Any surgical intervention of the knee
* Local or systemic infection
* Any patient with sever renal Impairment
* Bleeding disorders

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
knee osteoarthritis pain | six months following injection
  according to Visual Analogue Scale (VAS) which is a subjective scale used to quantitatively assess pain (0-10, 0 = No pain, 10 = Severe pain).
Decrease of Analgesic requirement for pain control after injection | six months following injection
  One week before injections all patients will be given etoricoxib 60 mg orally once daily and if pain is not controlled on this dose etoricoxib dose will be increased to 90 mg per day orally, if pain is still patient will add paracetamol 665 mg once daily orally up to 3 times per day till patient reach satisfactory level of pain control, analgesic type and dose will be recorded , patients will continue on these analgesia till the end of injection sessions , after injections the dose of analgesia will reduced gradually on opposite way till the patient reach the same satisfactory level of pain control before injection then the doses of analgesics will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ahmed Hamdy saied Ayad, Tanta, El-Gharbia
  - Tanta University, Tanta

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator
Supporting Information: Study Protocol
Time Frame: one year